CLINICAL TRIAL: NCT07063498
Title: The Effect of Fake Coughing and Stress Ball Application on Pain During Bone Marrow Aspiration and Biopsy
Brief Title: Fake Coughing During Bone Marrow Aspiration and Biopsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Gui Dural, PhD, Firat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/03-04
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-09

CONDITIONS: Bone Marrow Aspiration and Biopsy; Pain; Feigned Cough; Stress Ball
Keywords: bone marrow aspiration and biopsy; Pain; Stress
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cough Group (Experimental): Voluntary Coughing Maneuver
  Interventions: Behavioral: Coughing Maneuver
- control phase (No Intervention): Patients undergo biopsy without any additional intervention.
- Stress Ball Group (Experimental): Stress Ball Intervention
  Interventions: Behavioral: Stress ball

INTERVENTIONS:
Behavioral: Coughing Maneuver — 1. Voluntary Coughing Maneuver (Hileli Öksürük): Patients in this group were instructed to perform a voluntary coughing maneuver immediately prior to the percutaneous biopsy procedure. The maneuver was demonstrated by the clinician, and patients were asked to perform 2-3 forceful coughs while in the biopsy position, 30 seconds before needle insertion, to reduce anxiety and procedural pain perception.
  Arms: Cough Group
Behavioral: Stress ball — 2. Stress Ball Intervention: Patients were given a standard-sized rubber stress ball to hold and repeatedly squeeze during the entire percutaneous biopsy procedure. The intervention began 1 minute before needle insertion and continued until the procedure was completed. The aim was to provide a behavioral distraction to alleviate anxiety and pain.
  Arms: Stress Ball Group

SUMMARY:
Hematology patients go through many difficult periods during the diagnosis process. One of the most commonly used methods in the diagnosis of hematological diseases is bone marrow aspiration and biopsy (BMAB). BMAB is an invasive procedure and may cause pain in patients. For this purpose, a local anesthetic agent is used during the procedure. However, no effective method has been developed to prevent pain in patients. Both pharmacological and non-pharmacological methods are used to manage pain. Among non-pharmacological methods, cognitive distraction techniques such as feigned coughing and stress balls are used to reduce pain and stress. Some studies have reported that "fake coughing" reduces pain during procedures that cause temporary, sharp pain, such as parenteral injections or venipuncture. A literature review revealed that patients undergoing bone marrow aspiration and biopsy experience intense stress and pain, but there are insufficient studies examining these concepts. This study is expected to contribute to the nursing literature. The aim of this study is to determine the effect of fake coughing and stress ball application on pain during bone marrow aspiration and biopsy.

DETAILED DESCRIPTION:
Hematology patients go through many difficult periods during the diagnostic process. One of the most commonly used methods in the diagnosis of hematological diseases is bone marrow aspiration and biopsy (BMAB). BMAB is an important examination performed to reveal the cellular characteristics of the bone marrow and the involvement of solid organs or hematological malignancies when there is suspicion in peripheral blood. This procedure plays an important role in the diagnosis of primary and secondary malignant diseases as well as hematological diseases. It can also assist in the staging and sometimes diagnosis of lymphoproliferative diseases, the investigation of unexplained fever, and the diagnosis of disseminated fungal infections and storage diseases. Furthermore, bone marrow aspirations and biopsies have proven useful in detecting non-hematological malignancies in cases where malignancies are not clinically suspected. When both procedures are performed simultaneously, they complement each other, providing more material to examine the morphology and distribution pattern of cells. BMB can be performed in both inpatient and outpatient settings. The posterior iliac crest is the preferred and most common target site for KİAB due to its superficial location, technical ease, and the absence of critical structures along the needle path. The excellent safety profile and high diagnostic yield of KİAB have been established in the literature, making this intervention a critical component of patient management in contemporary medical practice.

Due to its invasive nature, KİAB may cause pain in patients. For this purpose, a local anesthetic agent is used during the procedure. However, no effective method has been developed to prevent pain in patients. In addition to pain, these patients may experience anxiety symptoms such as worry and uncertainty before the procedure. The literature acknowledges the lack of information on pain reduction during the KİAB procedure. Since the importance of more information in this area is recognized, there are no clear guidelines on how to use data on pain-causing factors to prevent or manage pain in patients undergoing this type of biopsy. Nevertheless, the limited studies conducted to reduce procedure-related pain have not changed clinical practice, and pain continues to be a significant burden for many hematological patients.

There are many independent factors that have been investigated in relation to pain in KİAB. These include gender, age, body mass index (BMI), educational level, pre-procedure knowledge, previous KİAB experience, KİAB indication, KİAB site, operator experience, duration, and procedure difficulty. When considering separate characteristics such as BMI, age, or operator experience, study results are often inconsistent. The correlation between procedure duration and difficulty and pain has been documented in various studies. Both pharmacological and non-pharmacological methods are used in pain management. Among non-pharmacological methods, cognitive distraction techniques such as feigned coughing and stress balls are used to reduce pain and stress.

Some studies have reported that "fake coughing" reduces pain during procedures that cause temporary, sharp pain, such as parenteral injections or venipuncture. In this technique, the patient is instructed to cough during the injection or venipuncture procedure. There are several theories about how this maneuver reduces pain, including distraction, stimulation of the autonomic nervous system (coughing has been theorized for this purpose), and increased pressure activating segmental pain-blocking pathways in the subarachnoid space .

It is noted that stress is a result of being unable to cope with emotional or physical threats, and that a person's mental health is closely and directly related to perceived stress. Although there are many methods for reducing stress, it is thought that a stress ball, which is inexpensive and easily accessible, can be used as a method of distracting or redirecting attention. The use of stress balls during minimally invasive venous surgery has been found to reduce anxiety and pain levels.

A literature review revealed that patients undergoing bone marrow aspiration and biopsy experience intense stress and pain, but there are insufficient studies examining these concepts. This study is expected to contribute to the nursing literature. The aim of this study is to determine the effect of feigned coughing and stress ball application on pain during bone marrow aspiration and biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer at least 3 months ago
* Over 18 years of age
* Able to communicate adequately
* No psychiatric problems
* Willing to participate in the study

Exclusion Criteria:

* Patients with communication problems
* Patients with psychiatric problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-22 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity During Bone Marrow Aspiration and Biopsy | Immediately after the procedure.
  Patient-reported pain intensity during bone marrow aspiration and biopsy procedures measured by a 10-point Visual Analog Scale (VAS), where 0 = no pain and 10 = worst pain imaginable.

IPD SHARING:
Plan to Share IPD: No